CLINICAL TRIAL: NCT05744258
Title: A Prospective Exploratory Study on the Value of Bio-electrical Impedance Analysis in Irritable Bowel Syndrome
Brief Title: The Value of Bio-electrical Impedance Analysis in Irritable Bowel Syndrome
Acronym: BIA-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BIA-IBS
Record Dates: First submitted 2023-01-27; First posted 2023-02-24 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS patients (Other)
  Interventions: Device: Bio-electrical impedance analysis
- Healthy volunteers (Other)
  Interventions: Device: Bio-electrical impedance analysis

INTERVENTIONS:
Device: Bio-electrical impedance analysis — Bio-electrical Impedance Analysis will be performed by trained personnel. BIA will be performed after fasting for at least 6 hours. Subjects should refrain from intensive physical activity the day be-fore the measurement. For women, measurements will be performed outside menstruating periods. Subjects will lay down on an examination couch with bare feet. Any jewelry will be removed.
  Reactance and resistance will be obtained. Phase angle will be calculated according to the formula:
  PhA (°) = (reactance/ resistance° x (180°/π). Body composition, including muscle mass and percentage body fat will be calculated.

SUMMARY:
The study aim is to investigate the Bio-electrical Impedance (BIA) parameters in general, and phase angle (PhA) in particular in Irritable bowel syndrome (IBS) patients and to compare these with values from healthy controls, while assessing the relationship with other confounding parameters in IBS: psychological parameters, physical activity, dietary pattern (with special interest in FODMAP intake). In a second phase, the evolution of the BIA parameters will be analyzed according to response to therapy.

DETAILED DESCRIPTION:
The role and significance of bio-electrical impedance analysis (BIA) has not been studied in IBS. Therefore, The investigators designed this exploratory study to assess its potential role in the diagnosis and follow-up of treatment in IBS. The study aim is to investigate the BIA parameters in general, and PhA in particular in IBS patients and to compare these with values from healthy controls, while assessing the relationship with other confounding parameters in IBS: psychological parameters, physical activity, dietary pattern (with special interest in FODMAP intake). In a second phase, the evolution of the BIA parameters will be analyzed according to response to therapy.

The primary objective is to compare the BIA parameters including PhA between IBS and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 75 years;
* Fulfilling the ROME IV criteria for IBS (only for patients);

Exclusion Criteria:

* Clinical suspicion of an organic disorder different from IBS (patients can be included when this disorder had been excluded);
* Known inflammatory bowel disorder;
* Known major intestinal motility disorder;
* Alcohol (defined as more than 14 U per week) or other substance abuse;
* Active psychiatric disorder;
* Known systemic or auto-immune disorder with implication for the GI system;
* Prior abdominal surgery (with the exception of cholecystectomy or ap-pendectomy);
* Any prior diagnosis of cancer other than basocellular carcinoma;
* Current chemotherapy;
* History of gastro-enteritis in the past 12 weeks;
* Dietary supplements unless taken at a stable dose for more than 12 weeks;
* Treatment with neuromodulators (one neuromodulator taken at a sta-ble dose for more than 12 weeks is allowed);
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our first patient was recruited on the 22nd of August 2022. The last patient entered the study on 15JUN2023. Patients with IBS were recruited at the gastro-enterology department. Healthy volunteers were asked to participate in the hospital.
Pre-assignment Details: Signing of the ICF, screening and baseline visit were all done on the same day. One patient withdrew consent and was excluded.
Groups:
- IBS Patients: patients having irritable bowel disease
- Healthy Volunteers: participants not having irritable bowel disease or bowel problems
Period: Overall Study
Arm/Group | IBS Patients | Healthy Volunteers
Started | 20 | 20
Completed | 16 | 20
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: patients not having irritable bowel disease or any bowel problems
- Total: Total of all reporting groups
Arm/Group | IBS Patients | Healthy Volunteers | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 35
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 2 | 11 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Median (Standard Deviation); unit: kg/m2] | 27.23 (6.46) | 23.77 (3.76) | 25.54 (5.11)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Phase Angle Between IBS Patients and Healthy Individuals
Description: Bio-electrical Impedance Analysis will be performed by trained personnel. BIA will be performed after fasting for at least 6 hours. Subjects should refrain from intensive physical activity the day be-fore the measurement. For women, measurements will be performed outside menstruating periods. Subjects will lay down on an examination couch with bare feet. Any jewelry will be removed.
  Reactance and resistance will be obtained. Phase angle will be calculated according to the formula:
  PhA (°) = (reactance/ resistance° x (180°/π).
Time Frame: The phase angle will be assessed through study completion, an average 6 months
Measure: Median (Standard Deviation); unit: degrees
Groups:
- IBS Patients: patients suffering from irritable bowel syndrome
- Healthy Volunteers: participants not suffering from irritable bowel syndrome
Arm/Group | IBS Patients | Healthy Volunteers
Number analyzed (Participants) | 16 | 20
degrees | 5.78 (0.53) | 6.35 (0.65)

2. Primary Outcome: Comparison of the Percentage of Total Body Water Between IBS Patients and Healthy Individuals
Description: percentage of total body water will be calculated using the measurements obtained during the BIA analysis.
Time Frame: The body composition will be assessed through study completion, an average 6 months
Measure: Median (Standard Deviation); unit: % of total body water
Groups:
- IBS Patients: patients suffering from IBS
- Healthy Volunteers: participants not suffering from IBS
Arm/Group | IBS Patients | Healthy Volunteers
Number analyzed (Participants) | 16 | 20
% of total body water | 63.4 (9.8) | 72.3 (7.8)

3. Primary Outcome: Comparison of the Muscle Mass Between IBS Patients and Healthy Individuals
Description: The muscle mass will be calculated using the measurements obtained during the BIA analysis.
Time Frame: the muscle mass will be assessed through study completion, an average 6 months
Measure: Median (Standard Deviation); unit: % of muscle mass
Arm/Group | IBS Patients | Healthy Volunteers
Number analyzed (Participants) | 16 | 20
% of muscle mass | 42.9 (6.39) | 52.6 (5.44)

4. Primary Outcome: Comparison of the Percentage of Body Fat Between IBS Patients and Healthy Individuals
Description: percentage of body fat will be calculated using the measurements obtained during the BIA analysis.
Time Frame: the percentage of body fat will be assessed through study completion, an average 6 months
Measure: Mean (Standard Deviation); unit: % of fat free mass
Groups:
- Healthy Volunteers: participants suffering from IBS
Arm/Group | IBS Patients | Healthy Volunteers
Number analyzed (Participants) | 16 | 20
% of fat free mass | 46.8 (6.8) | 53.7 (3.8)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow up, up to 1 week
Description: safety was checked for all patients, however every patient only performed 1 visit. They were followed until 1 week after that visit regarding safety but no AE's, SAE's or deaths occurred.
Groups:
- IBS Patients: participants suffering from IBS
Arm/Group | IBS Patients | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT05744258/Prot_SAP_000.pdf